CLINICAL TRIAL: NCT04646863
Title: Effect of Class IV Laser Therapy and Pilates Exercises on Bone Density and Pain in Primary Osteoporosis: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Emad Eldin Mohamed, Clinical Professor, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00400
Record Dates: First submitted 2020-11-21; First posted 2020-11-30 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, LLLT, multiwave locked system laser, Physical therapy modalities, DEXA, Pilates exercises
MeSH Terms: conditions — Osteoporosis | interventions — Laser Therapy; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): consists of 20 patients received a multiwave locked system laser
  Interventions: Radiation: laser therapy
- group B (Experimental): consists of 20 patients received Pilates exercises
  Interventions: Other: exercise
- group C (Experimental): consists of 20 patients received a multiwave locked system laser and Pilates exercises
  Interventions: Other: combination

INTERVENTIONS:
Radiation: laser therapy — performed by MLS® Laser Therapy (ASA Srl, Vicenza, Italy). It is designed to synchronize between two modules. One is emitting at 905 nm, with peak optical power = 25 W; each pulse is composed of a pulse train (single pulse width = 100 ns, maximum frequency 90 kHz). The frequency of the pulse trains varied between 1 and 2000 Hz. The other one is emitting at 808 nm in a continuous mode (power 1.1 W) or pulsed mode (pulses repetition rate 1-2000 Hz).
  Arms: group A
Other: exercise — The exercises were applied on a floor mat to achieve a full body workout with 10 repetitions for each exercise and rest for one minute before beginning the next exercise to avoid muscle fatigue as the following.
  1. Modified Hundred
  2. Modified Single Leg Stretch
  3. One Leg Circle
  4. Modified Scissors
  Arms: group B
Other: combination — laser therapy + Pilates exercises
  Arms: group C

SUMMARY:
the current study was to investigate the effect of class IV laser therapy and Pilates exercises on bone density in Osteoporosis.Sixty patients with osteoporosis (T-score values below -2.5) in lumbar spine with no evidence of vertebral compression fractures were recruited from October 6 University Hospital and Kaser El-aini Hospital, Cairo - Egypt from February 2019 to November 2019. Their age ranged from 40 to 60 years old. Patients with a history of tumors, ovariectomy, heart disease, renal failure, disc prolapse, or any trauma to the back area were excluded from the study

DETAILED DESCRIPTION:
They were allocated randomly into three groups: Group A consists of 20 patients received a multiwave locked system laser, group B consists of 20 patients received Pilates exercises and group C consists of 20 patients received a multiwave locked system laser and Pilates exercises. Patients with a history of tumors, ovariectomy, heart disease, renal failure, disc prolapse, or any trauma to the back area were excluded from the study. All patients who participated in the current study did not intake any medications to accelerate bone density like vitamin D or calcium. The randomization method was applied by asking each patient to choose a piece of paper that the (A), (B), or (C) letter was written. (A) considered the LLLT group, (B) considered the Pilates exercise group, while (C) considered the LLLT and Pilates exercises group. Both patients, the examiner, and therapist were blinded from the selection process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoporosis (T-score values below -2.5)

Exclusion Criteria:

* Patients with a history of tumors, ovariectomy, heart disease, renal failure, disc prolapse, or any trauma to the back area

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-09-22 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
DEXA | 8 weeks
  Model QDR-1000W, NORLAND; Hologic Inc., Waltham, Massachusetts, USA was used to measure bone mineral density (BMD) of the lumbar spine in mg/cm2.
Numeric pain rating scale (NPRS) | 8 weeks
  Pain intensity was measured by using NPRS which consists of an11-points numeric scale range from '0' representing 'no pain' to '10' representing 'the worst pain'. All patients were instructed to choose a number from 0 to 10 that describe their pain. The classification of pain intensity on the scale was: 0 indicate no pain, points from 1-3 indicate mild pain, points from 4-6 indicate moderate pain, and points from 7-10 indicate severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Bassam, Cairo, Egypt